CLINICAL TRIAL: NCT02412293
Title: Community-based Perinatal and Newborn Care in Gilgit District, Northern Areas, Pakistan: an AKU-AKHSP Collaboration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Aga Khan Health Services (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Professor, Aga Khan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: AKU-AKHSP
Record Dates: First submitted 2015-03-31; First posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Perinatal Problems; Still Births; Neonatal Deaths
Keywords: Perinatal; neonatal; newborn; mortality
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Health Education & Promotion: LHWs and CHWs will delivered the package via community awareness sessions and two one-to-one counselling sessions to pregnant women during third trimester and five newborn assessment visits in the neonatal period in intervention areas.
  Training of Health Workers: The LHWs and CHWs will receive trainings on IMNCI-based training package.
  Community Mobilization: For community mobilization and education, two types of tools will be used one group session by use of flip charts and group session by use of video.
  Interventions: Behavioral: Health Education & Promotion; Other: Training of Health Workers; Behavioral: Community Mobilization
- Control (No Intervention): Control areas will continue to receive the routine standard health services of governmental and non-governmental organizations in the area.

INTERVENTIONS:
Behavioral: Health Education & Promotion — Promotion of antenatal care, adequate nutrition, skilled delivery and healthy newborn care practices at household level.
  Arms: Intervention
Other: Training of Health Workers — Training of health workers on recognition of danger sign that warrant referral to health care service.
  Arms: Intervention
Behavioral: Community Mobilization — Community mobilization activities included formation of community health committees and creation of support for the uptake of the interventions.
  Arms: Intervention

SUMMARY:
There is limited evidence from community-based interventions to guide the development of effective maternal, perinatal and newborn care practices and services in developing countries. Investigators planned to evaluate the impact of a low-cost package of community-based interventions implemented through government sector lady health workers (LHWs) and community health workers (CHWs) of a NGO namely Aga Khan Health Services on perinatal and neonatal outcomes in a sub-population of the remote mountainous district of Gilgit, Northern Pakistan.

A community-based package for use by LHWs and CHWs geared towards prevention and promotion of maternal and newborn health practices and services will be developed based on formative research in the study district. The package will include promotion of antenatal care, adequate nutrition, skilled delivery and healthy newborn care practices at household level. The health workers will be trained in recognition of danger sign that warrant referral to health care service. LHWs and CHWs will delivered the package via community awareness sessions and two one-to-one counselling sessions to pregnant women during third trimester and five newborn assessment visits in the neonatal period. In addition to this, community mobilization activities included formation of CHCs and creation of support for the uptake of the interventions. Control areas will continue to receive the routine standard health services of governmental and non-governmental organizations in the area. The intervention areas will receive the intervention package in addition to the routine standard health services. Outcome measures will include changes in maternal and newborn-care practices and perinatal and neonatal mortality rates between the intervention and control areas.

DETAILED DESCRIPTION:
The World Health Organization estimates that globally over 9 million infants die annually before birth or in the first few weeks of life, and that the majority of these deaths occur in the neonatal period. The bulk of these deaths result from pregnancy or delivery associated complications, premature births, intrauterine growth retardation and infectious diseases.

There are over seven million perinatal deaths annually globally mostly in developing countries. Almost 4 million newborns suffer moderate to severe birth asphyxia, with at least 800,000 dying and probably a higher number developing sequel such as epilepsy, mental retardation, cerebral palsy and learning disabilities. A recent community based study in Zimbabwe, which audited perinatal mortality showed the commonest single cause was perinatal asphyxia and an avoidable factor was detected in 76% of cases. In another population based study in Bangladesh, which showed a perinatal mortality rate of 75 per 1000 births (37 stillbirths, 38 first week deaths), the major causes of early neonatal death were attributed to a small size at birth (54%), birth asphyxia (26%), and tetanus (8%). In Bangalore, South India a prospective hospital based study of 4572 births showed a perinatal mortality of 43/1000. Using the Wiggles worth's classification , 24% were considered due to birth asphyxia, even after exclusion of the premature group. Similarly a recent evaluation of a large hospital-based birth cohort for perinatal deaths in Karachi according to the Wiggles worth's criteria, indicated that almost 30% of all deaths were related to acute asphyxia.

Hypotheses

1. A concerted and coordinated community-based program of training first level primary care workers i.e. TBAs, LHWs, lady health visitors and rural health center physicians in the prevention, early recognition and management of common perinatal / neonatal problems will result in a significant reduction in perinatal and neonatal mortality in the Northern areas of Pakistan.
2. A coordinated program of community education and awareness in the importance of perinatal care, prevention and recognition of neonatal problems will lead to improved neonatal health, better recognition of neonatal problems and care-seeking behavior.
3. The strengthening of secondary care perinatal and newborn care and reproductive health services will lead to improved referral patterns for perinatal / neonatal problems with better outcome.
4. Increasing the community awareness of neonatal problems and training of first level primary care workers will result in better domiciliary management of neonatal problems.

Phase 1: Formative Research The objectives of this first phase of the study are as follows

1. Determination of preconditions for studying care seeking practices (referral system, availability of BHU staff, doctors, LHVs)
2. Focusing questions for formative research on care-seeking and causes of perinatal / neonatal morbidity / mortality by a modified perinatal / neonatal verbal autopsy)
3. Rapid anthropological assessment of care-seeking behavior
4. Illness Episode and Channel Survey
5. Analysis of results of formative research
6. Identification of desired behaviors and changes
7. Selection of behaviors for intervention and their potential acceptability
8. Acceptability of planned intervention(s) for families, communities and care providers and possible additional structural changes

This initial phase of formative research, will be conducted in the Hunza-Karimabad/Nagar/Gojal tehsils of the Gilgit District of the Northern areas. A combined methodology of KAP survey and verbal/social autopsy will be employed. These will include an in-depth evaluation of knowledge, attitude and practices of families and primary care givers (TBAs, LHWs, LHVs and BHU/RHC staff) with regards to

* Common causes of maternal morbidity in pregnancy
* Maternal nutrition and dietary patterns in pregnancy
* Determinants of care seeking behavior during pregnancy and labor

  * Domiciliary versus hospital births
  * Selection of care givers by families
  * Reasons for referral by primary care givers
* Perception and recognition of danger signs during child birth by families and care givers
* Immediate and early newborn care practices (colostrum and prelacteal feeding, breastfeeding, cord care, temperature regulation, swaddling, skin care etc).
* Concepts of early neonatal morbidity and health seeking behavior;

  * Risk factors for birth asphyxia and meconium aspiration
  * Low birth weight and temperature regulation
  * Neonatal infection (local and generalized)
  * Seizures or spasms
  * Respiratory problems
  * Jaundice
  * Feeding difficulty

Phase 2: Implementation phase

The overall objectives of this phase of the intervention are introduction and implementation of simple education and training materials for families and caregivers for community-based perinatal and newborn care by means of a phased introduction of the program in the area. In addition primary care givers in the target villages of the study area would receive training in stabilization and early referral of sick newborns for secondary care.

The intervention package, consisting of awareness creation about positive maternal and newborn health care practices at household level such as importance of; seeking antenatal care, adequate nutrition during pregnancy and lactation, skilled birth attendance, early initiation of breastfeeding, delayed bathing recognition of danger signs that warrant for early referrals, will be developed in collaboration with the Aga Khan Health Services, Pakistan. The practices will promote though community mobilization and education strategy that included formation of Community Health Committee (CHC) and group education sessions using flip charts and videos.

The LHWs and CHWs in the intervention areas will provide with enhanced trainings on causes of perinatal and newborn mortality and risky maternal and newborn care practices and expecting to transmit the knowledge to the families to avoid such practices. They will receive training in delivering the intervention package through standardized workshops including hands on practice on use of specific Information Education and Communication (IEC) materials developed for this purpose. The recently modified and simplified integrated management of neonatal and childhood illnesses (IMNCI) based system formed the basis of screening, recognition of danger signs and referral. The CHWs will deliver interventions in LHW uncovered areas within the intervention areas.

Control areas will continue to receive the routine services of governmental and non-governmental organizations in the area. But the public health care facilities of both intervention and control areas will receive similar competency based trainings in stabilization and early referral of sick newborns for secondary care.

The intervention Package The LHWs and CHWs will receive trainings on IMNCI-based training package. They will also receive orientation about the purpose of the project and how can they facilitate group education session by using flip charts and videos. The community-based health education sessions will be introduced targeting local communities to sensitize them regarding maternal, perinatal and newborn health issues.

In addition to this, Two days training workshops will be organized to train TBAs in intervention areas on "Clean Delivery Practices" at nearest health facilities. The UNICEF manual of (DAI) training will be adopted for this training.

The intervention package will be delivered through monthly household visits, one-to-one counseling sessions with pregnant women and video sessions in communities. Additionally, LHWs and CHWs in the intervention areas will record information about home visits, newborn illnesses, referrals, live births and deaths on special format designed for this project.

For community mobilization and education, two types of tools will be used one group session by use of flip charts and group session by use of video. Participants will be invited from all Muhallas (Sub-geographical distribution of the village population) to attend the session, facilitated by LHW/CHW to organize the session. Separate sessions will be organized for males and females. One session per area will be organized on quarterly basis in local school or LHW health house or CHW household within intervention areas. Target groups will be women of reproductive age, adolescent girls, fathers, mothers and fathers in law and mothers in law.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women & participants who agree to participate in the study

Exclusion Criteria:

* Pregnant women & participants who disagree to participate in the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3200 (Actual)
Dates: Start 2001-07; Primary Completion 2006-02 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Reduction in perinatal and neonatal mortality | 3 years
  Baseline & Endline Surveys

SECONDARY OUTCOMES:
Improvements in antenatal care practices | 3 Years
  Baseline & Endline Surveys
Improvements in cord application practices | 3 Years
  Baseline & Endline Surveys
Improvements in delaying first bath after birth | 3 Years
  Baseline & Endline Surveys
Improvements in colostrum administration | 3 Years
  Baseline & Endline Surveys
Improvements in initiation of breastfeeding practices within 1 hour after birth | 3 Years
  Baseline & Endline Surveys

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Result] Reducing Perinatal and Neonatal Mortality. Child Health Research Project Special Report. 1999;3:1-48.
- [Result] Costello AM. Perinatal health in developing countries. Trans R Soc Trop Med Hyg. 1993 Jan-Feb;87(1):1-2. doi: 10.1016/0035-9203(93)90395-7. PMID 8465375
- [Result] World Health Organization. Child health and development: health of the newborn. Geneva: World health Organization 1991.
- [Result] De Muylder X. Perinatal mortality audit in a Zimbabwean district. Paediatr Perinat Epidemiol. 1989 Jul;3(3):284-93. doi: 10.1111/j.1365-3016.1989.tb00380.x. PMID 2788880
- [Result] Fauveau V, Wojtyniak B, Mostafa G, Sarder AM, Chakraborty J. Perinatal mortality in Matlab, Bangladesh: a community-based study. Int J Epidemiol. 1990 Sep;19(3):606-12. doi: 10.1093/ije/19.3.606. PMID 2262255
- [Result] Wigglesworth JS. Monitoring perinatal mortality. A pathophysiological approach. Lancet. 1980 Sep 27;2(8196):684-6. doi: 10.1016/s0140-6736(80)92717-8. No abstract available. PMID 6106794
- [Result] Raghuveer G. Perinatal deaths: relevance of Wigglesworth's classification. Paediatr Perinat Epidemiol. 1992 Jan;6(1):45-50. doi: 10.1111/j.1365-3016.1992.tb00743.x. PMID 1553317
- [Result] Bhutta ZA. Perinatal care in Pakistan. Proceedings of the Symposium on Priorities in Perinatal Care in South Asia. September 1998, Karachi, Pakistan.
- [Derived] Memon ZA, Khan GN, Soofi SB, Baig IY, Bhutta ZA. Impact of a community-based perinatal and newborn preventive care package on perinatal and neonatal mortality in a remote mountainous district in Northern Pakistan. BMC Pregnancy Childbirth. 2015 Apr 30;15:106. doi: 10.1186/s12884-015-0538-8. PMID 25925407